CLINICAL TRIAL: NCT02778867
Title: Six Food vs One Food Eosinophilic Esophagitis Elimination Diet (SOFEED) Followed by Swallowed Glucocorticoid Trial
Brief Title: SOFEED: Six Food vs. One Food Eosinophilic Esophagitis Diet Study
Acronym: SOFEED
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Office of Rare Diseases (ORD) (NIH); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2015-1949; U54AI117804 (NIH)
Record Dates: First submitted 2015-10-12; First posted 2016-05-20 (Estimated); Results first posted 2020-05-26 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Eosinophilic Gastrointestinal Disorders (EGIDs); Eosinophilic Esophagitis (EoE)
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1-Food Elimination Diet (1FED) (Active Comparator): Participants eliminate milk from the diet in Phase 1
  Interventions: Other: 1 Food Elimination Diet Therapy
- 6-Food Elimination Diet (6FED) (Active Comparator): Participants eliminate milk, egg, wheat, soy, nuts, fish from the diet in Phase 1
  Interventions: Other: 6 Food Elimination Diet Therapy
- 1FED Non-Responders (6FED) (Other): Participants that fail to respond to 1FED in Phase 1 eliminate milk, egg, wheat, soy, nuts, fish from the diet in Phase 2
  Interventions: Other: 6 Food Elimination Diet (after 1FED failure)
- 6FED Non-responders (SGC) (Other): Participants that fail to respond to 6FED in Phase 1 administer swallowed glucocorticoids (SGC) (Flovent HFA) 880 mcg twice daily in Phase 2
  Interventions: Drug: Fluticasone Propionate, 880 mcg twice daily (after 6FED failure)

INTERVENTIONS:
Other: 1 Food Elimination Diet Therapy
  Arms: 1-Food Elimination Diet (1FED)
Other: 6 Food Elimination Diet Therapy
  Arms: 6-Food Elimination Diet (6FED)
Other: 6 Food Elimination Diet (after 1FED failure)
  Arms: 1FED Non-Responders (6FED)
Drug: Fluticasone Propionate, 880 mcg twice daily (after 6FED failure)
  Other Names: Flovent HFA
  Arms: 6FED Non-responders (SGC)

SUMMARY:
The purpose of this interventional study is to test and compare the effectiveness of two elimination diets-the 1-food elimination diet (1FED, milk only) and the 6-food elimination diet (6FED, milk, egg, wheat, soy, tree nut/peanuts, and fish/shellfish). The study will also test the effectiveness of swallowed glucocorticoid therapy in some of the study participants for whom diet therapy was not effective.

DETAILED DESCRIPTION:
This study will consist of two phases, plus a screening period. During the screening period, subject eligibility for the study will be determined. During Phase 1, qualified participants will be randomly assigned to one of two elimination diet therapies--the 1FED or the 6FED. Participants will remain on the assigned dietary therapy for 6 weeks. At the end of 6 weeks of therapy, esophageal biopsies from participant's standard of care (i.e. normal, routine care) endoscopy will be evaluated to determine disease status. Participants whose EoE is in remission (i.e. <15 eos/hpf) will be done with the study.

Participants whose EoE is still active (i.e. ≥15 eos/hpf) will have the option to continue into Phase 2 of the study. During Phase 2, participants who were on 1FED in Phase 1 will receive 6FED therapy for 6 weeks, and participants who were on 6FED during Phase 1 will receive swallowed glucocorticoid (SGC) therapy for 6 weeks. At the end of 6 weeks of therapy, esophageal biopsies from participant's standard of care (i.e. normal, routine care) endoscopy will be evaluated to determine disease status.

ELIGIBILITY:
Inclusion Criteria:

* Have diagnosis of EoE (based on consensus criteria)
* Have histologically confirmed active disease >15 eosinophils/hpf in either distal or proximal esophagus within 12 weeks of screening visit
* Symptomatic (have experienced symptoms within the last month prior to enrollment)
* Proton pump inhibitor (PPI) confirmation
* Have a negative urine pregnancy test at screening if of childbearing potential

Exclusion Criteria:

* Have been treated with topical swallowed steroids within the last 2 months or systemic steroids within the last 3 months
* Have pathological eosinophilia in segments of the GI tract other than the esophagus determined by local review
* Have been diagnosed with a GI malabsorption disorder (i.e., Inflammatory bowel disease, Crohn's disease) or Celiac disease
* Are currently on dietary therapy strictly avoiding milk or on a 6FED
* Have concurrent H pylori gastritis or parasitic infection
* Have history of anaphylaxis to milk (with current avoidance of milk)
* Have previously failed strict dietary therapy clearly documented with one of these regimens or topical steroid treatment (i.e. have achieved histological remission of <15 eos/hpf after having been on fluticasone or >1mg budesonide per day).
* Use of investigational drugs within 4 weeks (one month) prior to enrollment
* Are concurrently receiving any of the prohibited medications for the study
* On immunotherapy for pollen (if not on maintenance therapy) or immunoglobulin-E (IgE) -mediated food allergy
* Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2016-05-20 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc E Rothenberg, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (9):
- United States (9):
  - University of California, San Diego, La Jolla, California
  - Northwestern University, Chicago, Illinois
  - Tufts University, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina, Chapel Hill, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Kliewer KL, Gonsalves N, Dellon ES, Katzka DA, Abonia JP, Aceves SS, Arva NC, Besse JA, Bonis PA, Caldwell JM, Capocelli KE, Chehade M, Cianferoni A, Collins MH, Falk GW, Gupta SK, Hirano I, Krischer JP, Leung J, Martin LJ, Menard-Katcher P, Mukkada VA, Peterson KA, Shoda T, Rudman Spergel AK, Spergel JM, Yang GY, Zhang X, Furuta GT, Rothenberg ME. One-food versus six-food elimination diet therapy for the treatment of eosinophilic oesophagitis: a multicentre, randomised, open-label trial. Lancet Gastroenterol Hepatol. 2023 May;8(5):408-421. doi: 10.1016/S2468-1253(23)00012-2. Epub 2023 Feb 28. PMID 36863390
- See also: Consortium of Eosinophilic Gastrointestinal Disease Researchers — https://www.rarediseasesnetwork.org/cms/CEGIR

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from eosinophilic esophagitis specialty clinics (10 sites) in the USA between May 20, 2016 and March 2019
Pre-assignment Details: 143 participants screened, 14 excluded (8 did not meet inclusion criteria, 1 met exclusion criteria, 5 withdrew during screening), and 129 randomized
Groups:
- 1-Food Elimination Diet (1FED): Participants eliminate milk from the diet in Phase 1
  1 Food Elimination Diet Therapy
- 6-Food Elimination Diet (6FED): Participants eliminate milk, egg, wheat, soy, nuts, fish from the diet in Phase 1
  6 Food Elimination Diet Therapy
- 1FED Non-Responders (6FED): Participants that fail to respond to 1FED in Phase 1 eliminate milk, egg, wheat, soy, nuts, fish from the diet in Phase 2
  6 Food Elimination Diet Therapy
- 6FED Non-responders (SGC): Participants that fail to respond to 6FED in Phase 1 administer swallowed glucocorticoids (SGC) (Flovent HFA) 880 mcg twice daily in Phase 2
  Fluticasone Propionate, 880 mcg twice daily
Period: Phase 1
Arm/Group | 1-Food Elimination Diet (1FED) | 6-Food Elimination Diet (6FED) | 1FED Non-Responders (6FED) | 6FED Non-responders (SGC)
Started | 67 | 62 | 0 | 0
Completed | 65 | 59 | 0 | 0
Not Completed | 2 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 0 | 0
Period: Phase 2
Arm/Group | 1-Food Elimination Diet (1FED) | 6-Food Elimination Diet (6FED) | 1FED Non-Responders (6FED) | 6FED Non-responders (SGC)
Started | 0 (1FED non-responders from Phase 1 have the option to undergo 6FED in Phase 2) | 0 (6FED non-responders from Phase 1 have the option to undergo SGC in Phase 2) | 21 (Optional phase for 1FED non-responders) | 11 (Optional phase for 6FED non-responders)
Completed | 0 | 0 | 20 | 9
Not Completed | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1-Food Elimination Diet (1FED) | 6-Food Elimination Diet (6FED) | Total
Number analyzed (Participants) | 67 | 62 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (10.2) | 37.8 (10.4) | 37.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 29 | 59
  Male | 37 | 33 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 65 | 61 | 126
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 63 | 61 | 124
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 67 | 62 | 129
Peak Eosinophil Count [Median (Inter-Quartile Range); unit: eosinophils per high power field] — Maximum peak eosinophil count among distal, mid, and proximal esophageal biopsies Population: Clinical counts were used for study entry. Research counts (shown here) were unable to be obtained for some subjects.
  eosinophils per high power field
    number analyzed (Participants) | 64 | 59 | 123
    (all) | 56 [24 to 82] | 38 [25 to 61] | 44 [25 to 70]
Histology scoring system [Mean (Standard Deviation); unit: score on a scale] — The histology scoring system (HSS) measures the severity (grade) and extent (stage) of histologic abnormalities in the esophagus. Total score is the sum of grade and stage scores from the esophageal biopsy (distal, mid, or proximal) with the highest score (worst abnormalities) divided by the maximum possible score for the biopsy. Total scores range from 0 - 2 (higher scores indicate more severe and/or extensive abnormalities). Population: Histology scoring system scores were not obtained for some subjects at baseline (slides were unavailable)
  score on a scale
    number analyzed (Participants) | 64 | 59 | 123
    (all) | 0.83 (0.26) | 0.81 (0.25) | 0.82 (0.26)
Endoscopic Reference Score [Median (Inter-Quartile Range); unit: score on a scale] — The endoscopic reference score (EREFS) utilizes standardized criteria for the presence and degree of 5 major endoscopic features (edema, fixed rings, exudates, furrows, strictures). Total score is the sum of the five feature scores from the distal and proximal esophagus. Total scores range from 0 - 18 (higher scores indicate worsening features). Population: Baseline endoscopic feature scores were not obtained on some subjects
  score on a scale
    number analyzed (Participants) | 57 | 46 | 103
    (all) | 7.0 [4.0 to 9.0] | 6.5 [4.0 to 10.0] | 7.0 [4.0 to 10.0]

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants in Histologic Remission (<15 Eos/Hpf)
Description: Percent of participants in histologic remission in 1FED versus 6FED groups. Remission is defined as esophageal peak eosinophil count < 15 eosinophils per high powered field (eos/hpf)
Time Frame: 6 weeks after starting treatment
Population: Intent to treat analysis including participants who had at least one clinical observation post randomization. Participants whose histologic remission could not be determined were imputed as treatment failures.
Measure: Number; unit: percentage of participants
Arm/Group | 1-Food Elimination Diet (1FED) | 6-Food Elimination Diet (6FED)
Number analyzed (Participants) | 67 | 62
percentage of participants | 34.3 | 40.3
Statistical Analysis 1: Comparison: 1-Food Elimination Diet (1FED) vs 6-Food Elimination Diet (6FED); Test type: Other; p = 0.58, Fisher Exact — α < 0.05; Two-sided

2. Secondary Outcome: Percent of Participants in Complete and Partial Histologic Remission
Description: Percent of participants in complete and partial histologic remission in 1FED versus 6FED groups. Complete remission is defined as esophageal peak eosinophil count ≤ 1 eosinophils per high powered field (eos/hpf). Partial remission is defined as esophageal peak eosinophil count of 2 - 14 eos/hpf.
Time Frame: 6 weeks after starting treatment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 1-Food Elimination Diet (1FED) | 6-Food Elimination Diet (6FED)
Number analyzed (Participants) | 67 | 62
percentage of participants
  Complete remission (≤ 1eos/hpf) | 6.0 | 21.0
  Partial remission (2 - 14 eos/hpf) | 28.4 | 19.4
Statistical Analysis 1: Comparison: 1-Food Elimination Diet (1FED) vs 6-Food Elimination Diet (6FED); Test type: Other; p = 0.06, Fisher Exact — α < 0.05; Two sided

3. Secondary Outcome: Percent of Participants Following SGC in Histologic Remission in Phase 2
Description: Percent of participants who failed 6FED in Phase 1 in histologic remission after following swallowed glucocorticoids (SGC) in Phase 2. Remission is defined as esophageal peak eosinophil count < 15 eos/hpf
Time Frame: 6 weeks after starting treatment
Population: Intent to treat analysis including participants who had at least one clinical observation in Phase 2. Participants whose histologic remission could not be determined were imputed as treatment failures.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 6FED Non-responders (SGC): Participants that fail to respond to 6FED in Phase 1 administer swallowed glucocorticoids (Flovent HFA) 880 mcg twice daily in Phase 2
  Fluticasone Propionate, 880 mcg twice daily (after 6FED failure)
Arm/Group | 6FED Non-responders (SGC)
Number analyzed (Participants) | 11
percentage of participants | 81.8 [48.2 to 97.7]

4. Secondary Outcome: Percent of Participants Following 6FED in Histologic Remission in Phase 2
Description: Percent of participants who failed 1FED in Phase 1 in histologic remission after following 6FED in Phase 2. Remission is defined as esophageal peak eosinophil count < 15 eos/hpf
Time Frame: 6 weeks after starting treatment
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- 1FED Non-Responders (6FED): Participants that fail to respond to 1FED in Phase 1 eliminate milk, egg, wheat, soy, nuts, fish from the diet in Phase 2
  6 Food Elimination Diet (after 1FED failure)
Arm/Group | 1FED Non-Responders (6FED)
Number analyzed (Participants) | 21
percentage of participants | 42.9 [21.8 to 66.0]

5. Secondary Outcome: Change From Baseline in Peak Eosinophil Count
Description: Peak eosinophil counts were obtained at baseline and 6 weeks. The maximum (highest) peak eosinophil count among distal, mid, and proximal esophageal biopsies was obtained. Change in peak eosinophil count is defined as peak count at 6 weeks minus peak count at baseline. Changes in peak count are compared between 1FED and 6FED. A reduction (negative change) in peak count indicates improvement.
Time Frame: 6 weeks after starting treatment
Population: Intent to treat analysis including participants who had at least one clinical observation post randomization.
Measure: Median (Inter-Quartile Range); unit: eosinophils per high power field
Arm/Group | 1-Food Elimination Diet (1FED) | 6-Food Elimination Diet (6FED)
Number analyzed (Participants) | 64 | 59
eosinophils per high power field | -18 [-49 to 1] | -22 [-36 to -5]
Statistical Analysis 1: Comparison: 1-Food Elimination Diet (1FED) vs 6-Food Elimination Diet (6FED); Test type: Other; p = 0.90, Wilcoxon (Mann-Whitney) — α < 0.05

6. Secondary Outcome: Change From Baseline in Total Histology Scoring System
Description: The histology scoring system (HSS) measures the severity (grade) and extent (stage) of eight histologic abnormalities in the esophagus including eosinophilic inflammation, eosinophilic abscess, eosinophilic surface layering, surface epithelial alteration, dilated intercellular spaces, basal zone hyperplasia, dyskeratotic epithelial cells, and lamina propria fibrosis. Total score is the sum of grade and stage scores from the esophageal biopsy (distal, mid, or proximal) with the highest score (worst abnormalities) divided by the maximum possible score for the biopsy. Total scores range from 0 - 2 (higher scores indicate more severe and/or extensive abnormalities). Histology scores were obtained at baseline and 6 weeks. Change in total histology scoring system (HSS) is defined as total HSS score at 6 weeks minus total HSS score at baseline. Changes in scores are compared between 1FED and 6FED. A reduction (negative change) in score indicates improvement.
Time Frame: 6 weeks after starting treatment
Population: Intent to treat analysis including participants who had at least one clinical observation post randomization.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1-Food Elimination Diet (1FED) | 6-Food Elimination Diet (6FED)
Number analyzed (Participants) | 64 | 59
score on a scale | -0.15 (0.39) | -0.23 (0.34)
Statistical Analysis 1: Comparison: 1-Food Elimination Diet (1FED) vs 6-Food Elimination Diet (6FED); Test type: Other; p = 0.22, t-test, 2 sided — α < 0.05; Two sample t-test

7. Secondary Outcome: Change From Baseline in Total Endoscopic Reference Score
Description: The endoscopic reference score (EREFS) utilizes standardized criteria for the presence and degree of 5 major endoscopic features (edema, fixed rings, exudates, furrows, strictures). Total score is the sum of the five feature scores from the distal and proximal esophagus. Total scores range from 0 - 18 (higher scores indicate worsening features). Endoscopic features were assessed at baseline and 6 weeks. Change in total endoscopic reference score is defined as total score at 6 weeks minus total score at baseline. Changes in scores are compared between 1FED and 6FED. A reduction (negative change) in score indicates improvement.
Time Frame: 6 weeks after starting treatment
Population: Intent to treat analysis including participants who had at least one clinical observation post randomization.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 1-Food Elimination Diet (1FED) | 6-Food Elimination Diet (6FED)
Number analyzed (Participants) | 57 | 46
score on a scale | -1.0 [-4.0 to 0.0] | -2.0 [-4.0 to 1.0]
Statistical Analysis 1: Comparison: 1-Food Elimination Diet (1FED) vs 6-Food Elimination Diet (6FED); Test type: Other; p = 0.71, Wilcoxon (Mann-Whitney) — α < 0.05

ADVERSE EVENTS:
Time Frame: From informed consent to 30 days after the cessation of treatment
Groups:
- 6FED Non-responders (SGC): Participants that fail to respond to 6FED in Phase 1 administer swallowed glucocorticoids (SGC) (Flovent HFA) 880 mcg twice daily in Phase 2
  Fluticasone Propionate, 880 mcg twice daily (after 6FED failure)
Arm/Group | 1-Food Elimination Diet (1FED) | 6-Food Elimination Diet (6FED) | 1FED Non-Responders (6FED) | 6FED Non-responders (SGC)
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/62 | 0/21 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/62 | 0/21 | 1/11
Other Adverse Events (participants affected / at risk) | 1/67 | 2/62 | 0/21 | 4/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 1-Food Elimination Diet (1FED) (N=67) | 6-Food Elimination Diet (6FED) (N=62) | 1FED Non-Responders (6FED) (N=21) | 6FED Non-responders (SGC) (N=11)
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 1-Food Elimination Diet (1FED) (N=67) | 6-Food Elimination Diet (6FED) (N=62) | 1FED Non-Responders (6FED) (N=21) | 6FED Non-responders (SGC) (N=11)
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Bronchial Infection (Infections and infestations) | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (3):
  • Informed Consent Form (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/67/NCT02778867/ICF_000.pdf
  • Statistical Analysis Plan (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT02778867/SAP_001.pdf
  • Study Protocol (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT02778867/Prot_002.pdf